CLINICAL TRIAL: NCT06540638
Title: A Web-Based Education Program in Promoting Brain Health During the Surgical Journey in Older Patients
Brief Title: Cognitive Health Awareness Program in Surgical Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 24-5067
Record Dates: First submitted 2024-08-02; First posted 2024-08-06 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Dementia; Cognitive
Keywords: Educational Program; Cognitive Impairment; Postoperative Delirium
MeSH Terms: conditions — Dementia; Cognitive Dysfunction; Emergence Delirium

STUDY DESIGN:
Intervention Model Description: Single Group Assignment In a pre-operative assessment 1-30 days prior to their scheduled surgery, patients will be asked to participate in our web-based educational program. The program will be delivered on a research laptop/iPad at the clinic. The entire program, including pre- and post-education questionnaires and satisfaction survey should take about 20 minutes to complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- web-based education program (Experimental): Older surgical participants will receive a web-based educational program in promoting brain health (intervention). Participants will complete pre- and post-education questionnaires and a post-education satisfaction survey.
  Interventions: Behavioral: Web based education program

INTERVENTIONS:
Behavioral: Web based education program — In a pre-operative assessment, 1-30 days prior to their scheduled surgery, patients will be asked to participate in our web-based educational program. The content of our e-module included: introduction to brain health, surgery, and delirium, causes and risk factors, modifiable risk factors, and delirium prevention. The program will be delivered on a research laptop/iPad at the clinic. The entire program, including pre- and post-education questionnaires and satisfaction survey should take about 20 minutes to complete.

SUMMARY:
Addressing brain health and cognitive impairment (CI) in the aging population is important, especially in those undergoing surgery. While certain adverse outcomes are beyond control due to various factors, some may be preventable, such as delirium. It is crucial for patients and their families to be fully aware of the heightened risks associated with CI. By discussing the implications for individuals and their families, patients can make informed decisions about their health. Additionally, patients can be better prepared for their post-operative care and informed about post-operative complications. Education is a practical and viable solution to promote awareness and empower individuals to manage their cognitive health, especially in the context of surgery. Also, it can act as an early intervention. Thus, there is a need to proactively educate older adults about brain health.

The objective of the Web-Based Brain Health Education Study is to determine the impact of preoperative education on the knowledge of cognitive health of older surgical patients. Specifically, our study will examine the changes in knowledge scores after patients participate in a web-based education program on promoting brain health during their surgical journey. We hypothesize that a web-based education program will increase patient knowledge and empower them proactively about their brain health during the surgical journey.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the impact of a web-based educational program in promoting brain health in older surgical patients by changes in their knowledge score after education. For the secondary objectives, we aim to 1) determine participant satisfaction with the educational program, and 2) gain insights regarding perceived benefits and drawbacks of the brain health program.

This multicenter study will target older patients from pre-admission clinics at Toronto Western (TWH) and Mount Sinai Hospitals (MSH). Written informed consent to participate in the study will be obtained from all patients in person during the visit.

In a pre-operative assessment 1-30 days prior to their scheduled surgery, patients will be asked to participate in our web-based educational program. The program will be delivered on a research laptop/iPad/ paper version at the clinic. The entire program, including pre- and post-education questionnaires and satisfaction survey should take about 20 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

* patients ≥60 years old
* undergoing elective non-cardiac surgery
* competent to provide informed consent in English and
* possess some computer skills

Exclusion Criteria:

* previous major neurocognitive disorder
* uncontrolled psychiatric disorders
* hearing and/or vision impairment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in knowledge scores | At pre-surgery
  A knowledge questionnaire was developed to assess patient's knowledge of brain health during their surgical journey based on our education e-module. Our questionnaire contains 20 True/False questions. Each correct answer is worth one point, giving a minimum value/score of 0 and maximum value/score of 20. Higher values/scores indicate greater knowledge of brain health. The pre- and post-education questionnaires are identical.

SECONDARY OUTCOMES:
Participant satisfaction | At pre-surgery
  Participants will be asked to rate their level of satisfaction with the educational program.

CONTACTS AND LOCATIONS:
Overall Officials: Frances Chung, MBBS, FRCPC, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - 399 Bathurst St. Toronto Western Hospital, Preadmission Clinic, Dept. of Anesthesia, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No